CLINICAL TRIAL: NCT00860977
Title: VALacyclovir In Delaying Antiretroviral Treatment Entry
Brief Title: Can Valacyclovir Delay the Need for Initiation of Human Immunodeficiency Virus (HIV) Treatment in HIV-infected Individuals?
Acronym: VALIDATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN 240; ISRCTN66756285
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: HIV Infection; Herpes Simplex Type II; HIV Infections
Keywords: HIV; Herpes simplex virus type II; Genital herpes; Treatment Naive
MeSH Terms: conditions — HIV Infections; Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Odourless placebo tablet identical to valacyclovir in appearance and taste, to be taken twice daily
  Interventions: Drug: Placebo
- Valacyclovir (Experimental): oral valacyclovir 500mg twice daily
  Interventions: Drug: valacyclovir

INTERVENTIONS:
Drug: valacyclovir — oral valacyclovir 500mg twice daily
  Other Names: Valtrex
  Arms: Valacyclovir
Drug: Placebo — Odourless placebo tablet identical to valacyclovir in appearance and taste, to be taken twice daily
  Arms: Placebo

SUMMARY:
This study is a multicentre, randomized, placebo-controlled, fully blinded, clinical trial of twice daily oral valacyclovir 500mg versus placebo with the goal of delaying the need for initiating HAART among HIV infected individuals who neither use nor require HAART, and who have not used chronic suppressive anti-HSV therapy for at least the 6 months prior to study initiation.

ELIGIBILITY:
Inclusion Criteria:

* adult (aged 18 years or older or as per Local/Provincial Guidelines)
* documented HIV-1 infection (determined by EIA and Western blot, sites' standard assays are acceptable if approved in advance by the PIs for the study, Dr. Darrell Tan and/or Dr. Sharon Walmsley)
* no use of chronic anti-HSV therapy for the past 6 months, and not anticipated to require chronic anti-HSV therapy during the study
* antiretroviral naïve (no more than 14 days of total prior ARV exposure)
* CD4 count within the 400-900 cells/mm3 range (inclusive) on two consecutive occasions, with at least one measurement within 30 days of initiating trial (baseline visit)
* does not meet recommendations for initiating ARV therapy according to current guidelines

Exclusion Criteria:

* pregnancy or actively planning to become pregnant
* receiving chemotherapy, chronic steroid therapy or other immunomodulatory medications (e.g. interferon, azathioprine, methotrexate, TNF-alpha antagonists, etc.)
* Estimated creatinine clearance <30 mL/min
* Other medical condition likely to cause death within 24 months
* Enrolled in a therapeutic HIV vaccine or immunotherapy trial
* Enrolled in another trial investigating the impact of another intervention on HIV disease progression
* HIV elite controller (EC), phenotypically defined here as documented duration of HIV infection of ≥5 years, a persistent CD4 cell count ≥500 cells/mm3, and a persistent plasma HIV viral load of <1000 copies/mL in the absence of antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
annual rate of change in CD4 count, calculated as the slope of participants' CD4 count change / time. | up to 5 years

SECONDARY OUTCOMES:
time from baseline until reaching the composite of either a CD4 cell count ≤350 cells/mm3 measured on two consecutive occasions at least 1 month apart, or initiation of HAART for any reason, whichever occurs first. | up to 5 years
Annual rate of change in the CD4 cell count percentage, calculated as the slope of the participants' CD4 count percentage change over time | up to 5 years
Log10 plasma HIV viral load at 12, 24 and 36 months of follow-up | up to 5 years
Treatment-emergent adverse events and laboratory abnormalities (CBC, serum creatinine) | up to 5 years
Frequency of episodes of HSV reactivations at any anatomic site | up to 5 years
Proportion of microbiologically confirmed flares of HSV during the trial that are caused by laboratory-confirmed acyclovir-resistant HSV | up to 5 years
Overall quality of life as measured by the MOS-HIV questionnaire at each 6-monthly time point | up to 5 years

OTHER OUTCOMES:
analysis of inflammatory markers in HIV disease progression, HIV Resistance Mutations and other herpesvirus serologies | up to 6 years
genetic testing of HLA-B*5701 and HLA-B*5703 status, and future genetic markers related to HIV disease progression and the impact of herpes and valacyclovir | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walmsley, MD FRCPC MSc, Principal Investigator — University Health Network, Toronto; Darrell HS Tan, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (25):
- Fundación Huesped, Buenos Aires, Argentina
- Brazil (3):
  - Instituto de Pesquisa Clínica Evandro Chagas, Rio de Janeiro
  - Ambulatorio de Infectologia da UNIFESP, São Paulo
  - Centro de Referencia e Treinamento em DST/AIDS, São Paulo
- Canada (17):
  - University of Alberta, Edmonton, Alberta
  - B.C. Women's Hospital & Health Centre - Oak Tree Clinic, Vancouver, British Columbia
  - Vancouver Infectious Disease Clinic, Vancouver, British Columbia
  - Cool Aid Community Health Centre, Victoria, British Columbia
  - CDHA, QEII Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Health Sciences Centre, Hamilton, Ontario
  - The Ottawa Hospital, General Campus Divsions of Infectious Diseases, Ottawa, Ontario
  - University of Ottawa Health Services, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - St. Clair Medical Associates, Toronto, Ontario
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec-Pavillon CHUL, Québec
- United Kingdom (4):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - St. Stephen's AIDS Trust, London
  - St. Mary's Hospital, London

REFERENCES:
- [Background] Tan DH, Raboud JM, Kaul R, Grinsztejn B, Cahn P, Walmsley SL. Can herpes simplex virus type 2 suppression slow HIV disease progression: a study protocol for the VALacyclovir In Delaying Antiretroviral Treatment Entry (VALIDATE) trial. Trials. 2010 Nov 24;11:113. doi: 10.1186/1745-6215-11-113. PMID 21106086